CLINICAL TRIAL: NCT05894941
Title: Effects of Corrective Exercises and Postural Education on Forward Head Posture- A Randomized Controlled Trial
Brief Title: Effects of Corrective Exercises and Postural Education on Forward Head Posture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Forward Head Posture
Record Dates: First submitted 2023-05-11; First posted 2023-06-08 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Musculoskeletal Deformity
Keywords: Forward head Posture; Corrective Exercises; Postural Education; Craniovertebral and Shoulder angles; Posture; Musculoskeletal

STUDY DESIGN:
Intervention Model Description: The participants in each group will receive the same treatment throughout the trial
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All the participants will be randomly organized into 3 different groups by the researcher.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Corrective Exercises Group (Active Comparator): The researcher will teach a total of 6 evidence-based corrective exercises and stretches. The participants will perform this for the prescribed time for a minimum of 3 and 5 times a week for a total of 6 weeks of the trial.
  Interventions: Other: Corrective Exercises
- Postural Education Group (Active Comparator): Postural guidelines for doing daily activity especially sitting for prolonged periods and using electronic devices like computers and other electronic devices.
  Interventions: Other: Postural Education
- Control Group (No Intervention): This group will not receive either of the above mentioned treatments.

INTERVENTIONS:
Other: Corrective Exercises — A total of 6 evidence-based exercises and stretches namely; Upper trapezius stretch, Sternocleidomastoid stretch, pectoral stretch; Chin tuck exercise, YTWL exercise, and resisted/isometric neck extension exercise will be prescribed to the exercise group while the postural education group will follow the guidelines provided by National Institutes of Health (NIH) for using computers and other sources. The control group will receive no intervention.
  Arms: Corrective Exercises Group
Other: Postural Education — Postural guidelines for doing daily activity especially sitting for prolonged periods and using electronic devices like computers and other electronic devices.
  Arms: Postural Education Group

SUMMARY:
Forward head posture is one of the most common postural problems that we face today. Sitting for long periods in poor posture and the excessive use of electronic devices has become a high risk for this postural abnormality.

The goal of this [interventional study] is to [provide the participants with simple and easy corrective exercises for this abnormal posture which they can do anywhere at any time and to provide postural education and awareness on the matter.

DETAILED DESCRIPTION:
Forward head posture is one of the most common postural problems that we face today. Sitting for long periods in poor posture and the excessive use of electronic devices has become a high risk for this postural abnormality.

The goal of this [interventional study] is to [provide the participants with simple and easy corrective exercises for this abnormal posture which they can do anywhere at any time and to provide postural education and awareness on the matter. Also, this study aims in comparing both the treatment and education.] in [the people who have forward head posture or are more likely to develop it]. The main question[s] it aims to answer are:

* Does corrective exercises have any effect on improving forward head posture?
* Does postural education has any effect on improving forward head posture?

Participants in [-Exercise group will perform corrective exercises for 6 weeks

* Postural Education group will follow postural guidelines while doing daily tasks for 6 weeks
* Control group will do nothing in 6 weeks]. Researchers will compare [Corrective Exercise group with Postural Education group and control group] to see if [corrective exercise group or postural education group has any effect on forward head posture and compare the results with the control group].

ELIGIBILITY:
Inclusion Criteria:

1. Consent to participate in the study.
2. Young & Middle-aged Adults between the ages of 20-40 years
3. Craniovertebral angle less than or equal to 50°
4. Shoulder Angle less than or equal to 52°

Exclusion Criteria:

1. History of Trauma
2. Acute Neck Injuries e.g., Whiplash
3. Surgical history

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2023-05-12 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-10 (Actual)

PRIMARY OUTCOMES:
Craniovertebral Angle | 6 weeks
  The CVA is obtained by measuring the angle formed by the intersection of two lines drawn through particular anatomical landmarks and can be obtained using an image of the sagittal view of a person's head and neck. The first line is drawn from the tragus of the ear to the spinous process of the C7 vertebrae, and the second line is drawn through the spinous process of the C7 vertebrae horizontally. Although, there is no clear cut-off point threshold, identifying FHP for craniovertebral angle, in general, subjects with smaller craniovertebral angle i.e. less than 50 degrees have more Forward head posture
Shoulder Angle | 6 weeks
  It is considered as the angle between a horizontal line through the spinous process of the C7 vertebra and a line passes from the midpoint of the shoulder joint through the spinous process of the seventh cervical vertebra.

SECONDARY OUTCOMES:
Short Survey 36 Questionnaire | 6 weeks
  The 36-Item Short Form Survey (SF-36) is an outcome measure instrument that is often used, a well-researched, self-reported measure of health. The SF-36 is often used as a measure of a person or population's quality of life (QOL).
Numeric Pain Rating Scale | 6 weeks
  The Numeric Pain Rating Scale (NPRS) (an outcome measure) is a unidimensional measure of adult pain intensity. This 11-point numeric scale ranges from '0' representing one pain extreme (e.g., "no pain") to '10' representing the worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Ebru Akbuga, Principal Investigator — Assistant Professor
Locations (1):
- Yeditepe University, Istanbul, Atasehir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The participant data contains sensitive information like their contact and photographs. That is why this information will not be shared.

REFERENCES:
- [Background] Sheikhhoseini R, Shahrbanian S, Sayyadi P, O'Sullivan K. Effectiveness of Therapeutic Exercise on Forward Head Posture: A Systematic Review and Meta-analysis. J Manipulative Physiol Ther. 2018 Jul-Aug;41(6):530-539. doi: 10.1016/j.jmpt.2018.02.002. Epub 2018 Aug 11. PMID 30107937
- [Background] Ruivo RM, Pezarat-Correia P, Carita AI. Effects of a Resistance and Stretching Training Program on Forward Head and Protracted Shoulder Posture in Adolescents. J Manipulative Physiol Ther. 2017 Jan;40(1):1-10. doi: 10.1016/j.jmpt.2016.10.005. Epub 2016 Nov 11. PMID 27842938
- [Background] Heydari Z, Sheikhhoseini R, Shahrbanian S, Piri H. Establishing minimal clinically important difference for effectiveness of corrective exercises on craniovertebral and shoulder angles among students with forward head posture: a clinical trial study. BMC Pediatr. 2022 Apr 27;22(1):230. doi: 10.1186/s12887-022-03300-7. PMID 35477430